CLINICAL TRIAL: NCT03935464
Title: Pilot Trial to Examine the Feasibility, Acceptability and Impact of an Intervention Using a New Urine-based Tenofovir Adherence Assay
Brief Title: Point-of-care Urine Monitoring of Adherence: Testing a Real-Time Urine Assay of Tenofovir in PrEP
Acronym: PUMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kenya Medical Research Institute (Other); University of Washington (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AI143340; R01AI167699 (NIH); R01AI143340 (NIH)
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Risk Reduction
Keywords: PrEP, women, Kenya, adherence, POC monitoring, urine test,TDF, immunoassay
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Pilot Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): POC adherence testing by a urine TFV assay with feedback
  Interventions: Behavioral: PUMA
- Standard of Care (No Intervention): Follow Kenya's PrEP guidelines on standard adherence counselling

INTERVENTIONS:
Behavioral: PUMA — Collect urine on intervention participants and screen for presence of TFV. Feedback will be provided to the participant based on the results on their adherence with provision of standard adherence counseling.
  Arms: Intervention Arm

SUMMARY:
Worldwide expansion of pre-exposure prophylaxis (PrEP) with oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) will be critical to ending the HIV epidemic. However, maintaining daily adherence to PrEP can be difficult and the accuracy of self-reported adherence is often limited by social desirability bias. Pharmacologic adherence monitoring (measuring drug levels in a biomatrix) has been critical to the interpretation of the PrEP trials, but testing usually requires expensive equipment and skilled personnel. We have recently developed a point-of-care (POC) immunoassay to measure tenofovir in urine, allowing real-time adherence monitoring for the first time. We now want to test the acceptability, feasibility and preliminary impact of monitoring adherence in real-time using this novel POC assay with adherence feedback provided to the patient with supportive messaging (versus standard of care adherence counseling).

DETAILED DESCRIPTION:
The study is a pilot randomized trial to test the acceptability to participants, feasibility for providers, and impact on long-term metric of adherence among participants (assessed via tenofovir hair levels) of implementing a POC urine tenofovir test to provide real-time adherence feedback and enhanced adherence counseling among women on PrEP in Thika, Kenya. Eligible women (n=100) will be HIV-negative, ≥18 years old, and on PrEP. Participants will be randomized 1:1 to the intervention of providing real-time feedback via the urine assay versus standard-of-care adherence counseling. Acceptability will be assessed by a quantitative survey of participants at the end of the study, as well as by qualitative data collected via in-depth interviews (n=20) and focus group discussions (n=4 groups of 5-10 women each). Feasibility will be assessed by the proportion of women retained in the study, the mean number of missed visits, the proportion of planned urine assessments completed and messages delivered, while in-depth interviews with providers will explore the ease of administering the urine test. Tenofovir levels in hair serve as the long-term metric of adherence.

Feasibility outcome: The investigators will assess the feasibility of the intervention by interviewing health care providers, who will be administering this test at the clinical point of care in the future. The investigators will examine provider perceptions of the assay using in-depth interviews. These key informant interviews will be performed at the end of this study with the healthcare providers (up to 8) who delivered the counseling messages to intervention arm participants after performing the POC urine TFV test. The semi-structured interview guide will draw from the Unified Theory of Acceptance and Use of Technology (UTAUT) model.200 This model incorporates factors that influence technology acceptance (in this case, of the POC immunoassay): perceived usefulness (performance expectancy), complexity to use (effort expectancy), stigma/social harm (social influence), and benefits (facilitating PrEP adherence among patients). These interviews will also elicit barriers and facilitators to delivering the TFV assay-informed counseling messages.

Acceptability outcome: The investigators will conduct a mixed-methods assessment of the intervention arm participants' experiences with real-time monitoring and feedback at the end of the study. A quantitative survey and a qualitative interview guide for in-depth interviews of participants will draw from the Information-Motivation-Behavioral skills (IMB) model.205-212 Quantitative data collection will occur via standardized interviewer-administered questionnaires. Items to be assessed include the following: 1) Feelings about receiving their PrEP adherence results in real time; 2) Likelihood of participating in other studies using a similar design; 3) Likelihood of wanting to receive results of urine testing outside of a study while they are on PrEP; 4) Concern about the privacy and security of the data regarding their urine results; 5) Grading of the potential impact of knowing their urine TFV results on subsequent medication adherence; 6) Advantages and disadvantages of being told about their adherence in real time; 7) Likelihood of taking PrEP just before later study visits because they knew the urine test was being conducted; 8) Preferences regarding a yes/no assay versus an assay that provides information on "high", "moderate" or "low" adherence. A 5-point Likert item format will be used to assess graded items (such as the likelihood of wanting continued urine testing in the context of PrEP; feelings about the urine testing, ranging from negative to positive; concerns about privacy, ranging from low to high; the potential impact of real-time feedback on subsequent adherence, ranging from low to high). Other items (advantages and disadvantages of being told about adherence results) will provide pre-specified options with one "other" option for open-ended text fields.

Adherence outcome: A linear mixed effects linear regression model will estimate the effect of the intervention versus standard-of-care on logarithmically transformed levels of tenofovir in hair.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Adult, age ≥18 years old
* HIV-1 uninfected based on a negative HIV-1 rapid test
* Not currently enrolled in an HIV-1 prevention clinical trial
* Not currently in a sero-discordant relationship

  * Already taking PrEP and will be enrolled at the 3-month follow-up visit following PrEP initiation
  * Willing to be randomized to point-of-care tenofovir drug testing
  * Willing/able to provide informed consent to participate in the study
  * No contraindication to use of TDF or FTC
  * Note: Women who are pregnant or breast feeding at screening/enrollment are still eligible

Exclusion Criteria:

* HIV positive women
* under 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women 18 years and above who are HIV-negative on PrEP
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Gandhi, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- KEMRI Partners in Health and Research Development (PHRD), Thika, Thika, Near Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data in publicly accessible databases once study is complete and study findings disseminated.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 48 months from start of study
Access Criteria: Investigators conducting PrEP research.

REFERENCES:
- [Background] Gandhi M, Bacchetti P, Rodrigues WC, Spinelli M, Koss CA, Drain PK, Baeten JM, Mugo NR, Ngure K, Benet LZ, Okochi H, Wang G, Vincent M. Development and Validation of an Immunoassay for Tenofovir in Urine as a Real-Time Metric of Antiretroviral Adherence. EClinicalMedicine. 2018 Aug-Sep;2-3:22-28. doi: 10.1016/j.eclinm.2018.08.004. Epub 2018 Aug 31. PMID 30906930
- [Background] Gandhi M, Bacchetti P, Spinelli MA, Okochi H, Baeten JM, Siriprakaisil O, Klinbuayaem V, Rodrigues WC, Wang G, Vincent M, Cressey TR, Drain PK. Brief Report: Validation of a Urine Tenofovir Immunoassay for Adherence Monitoring to PrEP and ART and Establishing the Cutoff for a Point-of-Care Test. J Acquir Immune Defic Syndr. 2019 May 1;81(1):72-77. doi: 10.1097/QAI.0000000000001971. PMID 30664078
- [Background] Spinelli MA, Glidden DV, Rodrigues WC, Wang G, Vincent M, Okochi H, Kuncze K, Mehrotra M, Defechereux P, Buchbinder SP, Grant RM, Gandhi M. Low tenofovir level in urine by a novel immunoassay is associated with seroconversion in a preexposure prophylaxis demonstration project. AIDS. 2019 Apr 1;33(5):867-872. doi: 10.1097/QAD.0000000000002135. PMID 30649051
- [Derived] Okello P, Velloza J, Ogello V, Owidi E, Mogere P, Gakuo S, Chakravarty D, Biwott C, Chatterjee P, Mugo N, Gandhi M, Ngure K. Acceptability and feasibility of a urine-based tenofovir adherence assay for monitoring and providing feedback on PrEP adherence in Kenya. AIDS Care. 2025 Feb;37(2):324-336. doi: 10.1080/09540121.2024.2444556. Epub 2024 Dec 28. PMID 39733245
- [Derived] Gandhi M, Glidden DV, Chakravarty D, Wang G, Biwott C, Mogere P, Maina G, Njeru I, Kiptinness C, Okello P, Spinelli MA, Chatterjee P, Velloza J, Ogello V, Medina-Marino A, Okochi H, Mugo NR, Ngure K. Impact of a point-of-care urine tenofovir assay on adherence to HIV pre-exposure prophylaxis among women in Kenya: a randomised pilot trial. Lancet HIV. 2024 Aug;11(8):e522-e530. doi: 10.1016/S2352-3018(24)00125-5. Epub 2024 Jul 5. PMID 38976993
- [Derived] Drain P, Ngure K, Mugo N, Spinelli M, Chatterjee P, Bacchetti P, Glidden D, Baeten J, Gandhi M. Testing a Real-Time Tenofovir Urine Adherence Assay for Monitoring and Providing Feedback to Preexposure Prophylaxis in Kenya (PUMA): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2020 Apr 2;9(4):e15029. doi: 10.2196/15029. PMID 32238341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the Kenya Medical Research Institute (KEMRI) Partners in Health and Research Development (PHRD) clinical research center at Thika. This center is associated with 5 five community sites from which participants were recruited for the study including surrounding voluntary counselling and testing centers, churches, and community organizations. Participants on PrEP for the last 3 months were recruited. Study began recruiting from March 1, 2021.
Pre-assignment Details: 105 women were assessed for eligibility and 5 were found ineligible because 4 were unavailable for study procedures and 1 was underage. 100 participants were enrolled and 49 were assigned to urine test counselling and 51 assigned to standard of care procedures.
Period: Overall Study
Arm/Group | Intervention Arm | Standard of Care
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Standard of Care | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 51 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.3 (10.6) | 33.8 (8.2) | 33.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 51 | 100
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 49 | 51 | 100
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Long-term Adherence Metrics Via Hair Concentrations of Tenofovir and Short-term Adherence Metric of Urine Concentrations of Tenofovir.
Description: Primary outcome is number of participants in each arm with detectable hair concentrations of Tenofovir indicating long-term adherence at 12 months (undetectable levels defined long-term non-adherence), as well as urine concentrations of Tenofovir at 12 months as a short-term adherence metric.
Time Frame: 12 months for each participant from the time of enrollment
Population: Adult women not in sero-discordant partnerships were enrolled 3 months after PrEP initiation at the Kenya Medical Research Institute.
Measure: Count of Participants; unit: Participants
Groups:
- PUMA Intervention Arm: Point-of-care (POC) adherence testing by a urine TFV assay with feedback
  Collect urine on intervention participants and screen for presence of TFV. Feedback will be provided to the participant based on the results on their adherence along with provision of standard adherence counseling.
- PUMA Standard of Care: Follow Kenya's PrEP guidelines on standard adherence counselling
Arm/Group | PUMA Intervention Arm | PUMA Standard of Care
Number analyzed (Participants) | 49 | 51
Participants
  Detectable Tenofovir in hair indicating long-term adherence: number analyzed (Participants) | 42 | 41
  Detectable Tenofovir in hair indicating long-term adherence | 33 | 26
  Detectable Tenofovir in urine indicating short-term adherence: number analyzed (Participants) | 43 | 42
  Detectable Tenofovir in urine indicating short-term adherence | 31 | 19

2. Secondary Outcome: Feasibility Among Healthcare Providers of Providing Test Feedback to Participants
Description: Themes among PrEP providers about feasibility of providing urine assay feedback to study participants on PrEP. The In-depth interviews and focus group discussions were cross-sectional.
Time Frame: Completed after the participants' 12-month follow-up visit
Population: Healthcare providers who provide PrEP
Measure: Count of Participants; unit: Participants
Groups:
- Healthcare Providers: We conducted in-depth interviews with purposively-sampled healthcare providers (HCPs) who administered the urine assay.
Arm/Group | Healthcare Providers
Number analyzed (Participants) | 8
Participants
  Easy to Use | 6
  Feasible within routine care | 8
  Concerned about added workload | 3

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Intervention Arm | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51

LIMITATIONS AND CAVEATS:
As a result of the COVID-19 pandemic and associated lockdowns, protocol deviations occurred - specifically, dried blood spots were not collected for additional adherence monitoring and hair was only collected at 12 months. Further, the study had a relatively small sample size of 100 participants. Finally, the study results cannot be generalized to other populations on PrEP such as men.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT03935464/Prot_SAP_ICF_000.pdf